CLINICAL TRIAL: NCT03461809
Title: A Retrospective Study to Investigate the Efficacy and Relative Factors of Ocular Acupuncture in Ocular Motor Nerve Palsy Patients
Brief Title: A Retrospective Study of the Effects of Ocular Acupuncture on Ocular Motor Nerve Palsy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 20180204
Record Dates: First submitted 2018-02-04; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Oculomotor Nerve Palsy; Trochlear Nerve Palsy; Abducens Nerve Paralysis
Keywords: diplopia; ocular motor nerve palsy; acupuncture
MeSH Terms: conditions — Oculomotor Nerve Diseases; Trochlear Nerve Diseases; Abducens Nerve Diseases; Diplopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ocular motor nerve palsy treated by ocular acupuncture: Ocular motor nerve palsy patients who received ocular acupuncture treatment
  Interventions: Other: Ocular acupuncture

INTERVENTIONS:
Other: Ocular acupuncture — Patient's skin located in the extraocular muscles projection area is routinely disinfected. A diameter of 0.20 mm and length of 25 mm needle is inserted slowly. Piercing depth is about 20mm. The electropuncture apparatus is used, each group of electrodes are distinguished with different colors of wires to generate current stimulations of current 1.0~1.5 milliampere (mA), voltage 9 volt(V), frequency 1.5 hertz (Hz), and duration of 40 minutes.

SUMMARY:
This retrospective observational study is designed to assess the response to treatment with ocular acupuncture and its relative factors, in terms of diplopia status, ocular motility differences, and clinical features, in ocular motor nerve palsy patients. During this study, a retrospective data collection will be carried out using the information contained in the medical record of aimed patients, provided that the treatment with ocular acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Patient who received at lease 1 times of ocular acupuncture treatment
* Patient who received full set of ophthalmology & neurology assessment pre- and post-treatment.

Exclusion Criteria:

* patient who combined with extraocular muscles diseases, eg.thyroid eye disease
* patient who underwent periocular surgery
* patient who combined with congenital ocular motor nerve palsy, eg. Brown syndrome.
* patient who had untreated condition which may lead to ocular motor nerve palsy such as intracranial aneurysm and brain tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with ocular motor nerve palsy who received ocular acupuncture.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2018-03-15 (Estimated); Primary Completion 2018-05-15 (Estimated); Study Completion 2018-05-15 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy rate (Cure, Effective and Invalid) | Through study completion, an average of 1 month.
  Clinical efficacy rate (Cure, Effective and Invalid) assessed by investigator's discretion. Efficacy rate is calculated as number of patients with Cure and effective proportional to number of all cases.

SECONDARY OUTCOMES:
Diplopia angle | Through study completion, an average of 2 weeks.
  Patient's diplopia angle obtained by retrospective chart review.
Eyeball movement distance | Through study completion, an average of 2 weeks.
  Patient's eyeball movement distance obtained by retrospective chart review.
Distance between upper and lower eyelid. | Through study completion, an average of 2 weeks.
  Patient's distance between upper and lower eyelid obtained by retrospective chart review.

IPD SHARING:
Plan to Share IPD: Undecided